CLINICAL TRIAL: NCT06793618
Title: Effectiveness of the Z-Track Technique As a Pain-Reducing Strategy for Neonates During Intramuscular Injection: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Haider Jumaa Kareem, Academic Nurse, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NO. 37/ 2024
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Intramuscular Injection; Neonates; Neonatal Pain
Keywords: Pain; non-pharmacological pain managment
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: A randomized control trial with one intervention and one control group. post-test only
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Z-track technique (Active Comparator): To perform the zeta-track technique: In this method, the neonates are in supine position, the skin is moved and held from the injection site 2 to 3 cm to the side or downward using the non- dominant hand, to ensure that blood vessel wasn't penetrated aspiration on the syringe must perceive the injection and then the medication is to be injected slowly. Researcher assistant that is unaware of the injection method performs the recording of the pain intensity and leakage diameter on the observation form.
  Interventions: Other: Z-track technique
- Control group (No Intervention): the neonates receive the intramuscular injection using the conventional method and protocol used in the postnatal ward without any interventions

INTERVENTIONS:
Other: Z-track technique — In this method, the neonates are in supine position, the skin is moved and held from the injection site 2 to 3 cm to the side or downward using the non- dominant hand, to ensure that blood vessel wasn't penetrated aspiration on the syringe must perceive the injection and then the medication is to be injected slowly. Researcher assistant that is unaware of the injection method performs the recording of the pain intensity and leakage diameter on the observation form.
  Arms: Z-track technique

SUMMARY:
A quantitative study, true experimental, posttest-only design has been used for the current study. one intervention (the Z-track technique) and one control group involved in the study. The primary outcome measure is the Neonatal/Infant Pain Scale to be used immediately after intramuscular injections to measure the pain level among neonates.

ELIGIBILITY:
Inclusion Criteria:

* Neonates delivered through cesarean section
* Apgar score of 8 or more
* Weight between 2500 - 3500 grams
* neonates receiving IM injections
* Males / females
* term neonates between 37th and 42nd week of gestation

Exclusion Criteria:

* Congenital anomalies
* neonates who received intramuscular injection such as the Hepatitis B vaccine
* Low birth weight
* Preterms
* Neural tube defects
* neonates who are of normal vaginal delivery

Ages: 5 Minutes to 2 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 147 (Actual)
Dates: Start 2024-11-24 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2024-12-28 (Actual)

PRIMARY OUTCOMES:
Neonatal/ Infant Pain Scale | from the process of enrollment at the post-natal ward until the IM injection is administered (usually takes less than 1 hour)
  A scale developed specifically for newborn infants. Consists of 6 criterion (Face Expression, cry, Patterns of Breathing, leg and arm movements, Arousal status) Recommended for children less than 1 year old.

CONTACTS AND LOCATIONS:
Locations (1):
- Feminine and Children Educational Hospital, Samawah, Muthanna Governorate, Iraq

IPD SHARING:
Plan to Share IPD: No